CLINICAL TRIAL: NCT04008225
Title: Study of the Effects of Bronchoalveolar Lavage Liquid in the ARDS on the Functioning of the Neutrophil Polynuclear System
Acronym: BALARDS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_9885
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: ARDS, Human
Keywords: Bronchoalveolar lavage
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARDS group: Inpatients hospitalized in medical intensive care with a table of ARDS defined according to the Berlin criteria and requiring an BAL for a diagnostic purpose under a suspicion of pneumopathy acquired under mechanical ventilation.
  Interventions: Procedure: Bronchoalveolar lavage
- Control group: The control group will be made up of patients with an BAL considered normal (endoscopy patients from the pneumology department). The normality of the BAL is defined by a normocellular wash with cellularity: < 150,000 to 200,000 cells/mL Cell composition (formula): macrophages: 80-90%, lymphocytes 5 to 10% (< 20%), neutrophils: < 5%, eosinophils: < 2%.
  Interventions: Procedure: Bronchoalveolar lavage

INTERVENTIONS:
Procedure: Bronchoalveolar lavage

SUMMARY:
Firstly, the study assesses the effect of bronchoalveolar lavage fluid (BAL) from patients in (acute respiratory distress syndrome (ARDS) on the life span of PNNs and on the phagocytosis of apoptotic cells by macrophages and polynuclear neutrophil (PNN).

Then, the effect of an antibody directed against "high-mobility group box 1" protein (HMGB1) and the effect of metformin on efferocytosis are studied.

DETAILED DESCRIPTION:
ARDS (acute respiratory distress syndrome) is a syndrome that causes significant mortality and morbidity. This syndrome is characterized by an alveolitis with polynuclear neutrophil (PNN). PNNs play an important role in the persistence and in injuries induced by ARDS. Several animal studies have shown that lesional edema can be increased by two important mechanisms: the increase in the lifespan of PNNs in the lung and the decrease in the phagocytosis capacities of apoptotic cells (efferocytosis) by macrophages and PNNs.

However, confirmation of these data in humans does not exist, and knowledge of the mechanisms that may increase lung damage during ARDS will limit it and thus reduce the mechanical ventilation time of these patients as well as the mortality associated with ARDS.

" high-mobility group box 1 " (HMGB1) protein may be involved in reducing efferocytosis capacity. Similarly, activation of AMP-activated protein kinase (AMPk) could restore the clearance capacity of apoptotic cells in macrophages and PNNs.

ELIGIBILITY:
Inclusion Criteria:

* ARDS Group : Inpatients hospitalized in medical intensive care with an ARDS defined according to the Berlin criteria and requiring an BAL(for diagnostic purpose in suspicion of pneumopathy acquired under mechanical ventilation).
* Control group : The control population is made up with patients with a BAL considered normal (endoscopy patients from the pneumology department). The normality of the BAL is defined by a normocellular wash with cellularity: < 150,000 to 200,000 cells/mL Cell composition (formula): macrophages: 80-90%, lymphocytes 5 to 10% (< 20%), neutrophils: < 5%, eosinophils: < 2%.

Exclusion Criteria:

* Age < 18 years;
* Pregnant women ;
* Persons deprived of their liberty by judicial or administrative decision;
* Persons legally incapable;
* Persons not affiliated to a social security system;
* Previously immunocompromised patients (HIV infection, hematopathy, organ transplantation, immunosuppression);
* Patients who do not require a lung sample.

Age Groups: Child, Adult, Older Adult
Study Population: * ARDS Group : Inpatients hospitalized in medical intensive care with an ARDS defined according to the Berlin criteria and requiring an BAL(for diagnostic purpose in suspicion of pneumopathy acquired under mechanical ventilation).
  * Control group : The control population is made up with patients with a BAL considered normal (endoscopy patients from the pneumology department). The normality of the BAL is defined by a normocellular wash with cellularity: < 150,000 to 200,000 cells/mL Cell composition (formula): macrophages: 80-90%, lymphocytes 5 to 10% (< 20%), neutrophils: < 5%, eosinophils: < 2%.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Lifespan of the PNNs | 24 hours after BAL
  The lifespan of the PNNs is an indicator of apoptosis : two groups are compared with and without incubation in BAL fluid.
  Neutrophil necrosis was assessed by flow cytometry using a phycoerythrin-conjugated active caspase-3 apoptosis kit (Becton Dickinson, USA)

SECONDARY OUTCOMES:
PNNs phagocytic index | 24 hours after BAL
  This index relates the ability of the PNNs to produce neutrophil extracellular traps (NETs).
  The release of NETs was quantified by measuring fluorescence with a microplate fluorescence reader (Varioskan, ThermoFisher Scientific, USA).
Efferocytosis index | 24 hours after BAL
  The efferocytosis index was determined on 300 cells as the percentage of Human monocyte-derived macrophages (HMDMs) containing at least one ingested apoptotic neutrophil.
Increase of PNNs phagocytic index with HMGB1 activator | 24 hours after BAL
  PNNs phagocytic index is measured after incubation with an anti-HMGB1 neutralising antibody
Increase of Efferocytosis index metformin | 24 hours after BAL
  efferocytosis index was determined after incubation with an AMP-activated protein kinase (AMPK) activator (metformin)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TADIE, MD, PhD, Principal Investigator — University Hospital of Rennes
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No